CLINICAL TRIAL: NCT04997642
Title: Parkinson's Disease and Movement Disorders Clinical Database
Status: Recruiting | Type: Observational
Sponsor: University of Pennsylvania (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Daniel Weintraub, Professor of Psychiatry and Neurology, University of Pennsylvania
Other Study IDs: 820710; NIA U19 (Other: NIA)
Record Dates: First submitted 2021-08-01; First posted 2021-08-09 (Actual); Last update posted 2025-10-07 (Actual); Status verified 2025-10

CONDITIONS: Parkinson Disease; Parkinson Disease Dementia; Lewy Body Parkinson Disease; Lewy Body Dementia With Behavioral Disturbance
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 15 Years
Biospecimen Retention: Samples With DNA — Plasma and cerebrospinal fluid obtained with patient's consent. Biological samples including blood and spinal fluid may be collected from each database participant. Each participant will be given the option of allowing the collection of none, some, or both of the biological samples. Samples will be stored in a secure facility at the University of Pennsylvania Department of Pathology and Laboratory Medicine. If the subject consents, approximately 20 ml (4 teaspoons) of blood will be collected, and 25 ml (2 tablespoons) of spinal fluid will be collected.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Behavioral: neuropsychiatric and cognitive testing questionnaires — Demographic data such as race, sex, age Family History Risk Factor Questionnaire Hoehn and Yahr Stage UPDRS Parkinson's symptom checklist Medication list Neuropsychological Test Battery Behavioral Exams
  * Geriatric Depression Scale Quality of Life Questionnaire
  * PDQ-39, SF-12

SUMMARY:
The research database contains demographic and family history information, longitudinal information on the clinical symptoms, neuropsychological profile and treatments, stored biological samples, and brain images of patients with Parkinson's disease and related disorders receiving care at the Parkinson's disease and Movement Disorders Center and the Hospital of the University of Pennsylvania.

DETAILED DESCRIPTION:
The research database contains demographic and family history information, longitudinal information on the clinical symptoms, neuropsychological profile and treatments, stored biological samples, and brain images of patients with Parkinson's disease and related disorders receiving care at the Parkinson's disease and Movement Disorders Center (PDMDC) and the Hospital of the University of Pennsylvania.

The purpose of the research database is to have a comprehensive source of data that can be used for educational, research and patient care projects at the PDMDC. These data may be used for any study examining the relationship between treatment and clinical symptoms of patients with PD and related disorders. The main uses of the data are to:

* Determine the long term effects of Parkinson's disease and related conditions, including predictors of its motor and non-motor symptoms
* Identify genetic and other neurobiological factors related to the risk of developing Parkinson's disease and related disorders and their course
* Improve our understanding of how best to identify, diagnose, and manage motor and non-motor symptoms of Parkinson's disease and related conditions Evaluate biological markers of disease or response to therapy
* Identify patients who may be candidates for participation in trials of new medications.
* Identify patients who may be interested in participating in educational or developmental activities

Participants are seen annually for the first 4 years, biennially thereafter. The participants continue in the study until study end, withdrawal, or death on study.

ELIGIBILITY:
Inclusion Criteria:

Any person who receives medical care for the diagnosis of Parkinson's disease with mild cognitive impairment (MCI) or dementia may be eligible to participate in the research database. There are no limitations for database participation based on age, disease severity or presence of cognitive impairments, as long as the person is able to complete the research assessments.

Exclusion Criteria:

Absence of Parkinson's disease diagnosis. There are no limitations for database participation based on age, disease severity or presence of cognitive impairments, as long as the person is able to complete the research assessments.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Population will be derived from outpatient clinics, support groups, self-referral, and community members.
Sampling Method: Non-Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2019-09-30 (Actual); Primary Completion 2029-09-15 (Estimated); Study Completion 2029-09-15 (Estimated)

PRIMARY OUTCOMES:
Long term effects of Parkinson's disease | 5 years
  Determine the long term effects of Parkinson's disease and related conditions, including predictors of its motor and non-motor symptoms
Genetic and Neurobiological factors | 5 years
  Identify genetic and other neurobiological factors related to the risk of developing Parkinson's disease and related disorders and their course

SECONDARY OUTCOMES:
Identification and Diagnosis of Parkinson's disease | 5 years
  Improve our understanding of how best to identify, diagnose, and manage motor and non-motor symptoms of Parkinson's disease and related conditions

CONTACTS AND LOCATIONS:
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
The data in the research database are available to researchers both within the PDMDC and other researchers at the University and at other Institutions.
  Any release of data outside the PDMDC will be reviewed by the Principal Investigator and the Director of the PDMDC to ensure that the study is scientifically sound, that the research projects are covered by the subject's informed consent, and are compliant with HIPAA regulations. Once the study has been approved, a de-identified data extract is prepared and the data necessary to conduct the study are extracted from the database.
Supporting Information: Study Protocol, ICF